CLINICAL TRIAL: NCT04742842
Title: A Phase I, Double-blind, Dose-ranging, Randomised, Placebo-controlled Trial to Study the Safety and Immunogenicity of a DNA-based Vaccine Against COVID-19 (COVIGEN) in Healthy Participants Aged 18 to 75 Years Old
Brief Title: The Safety and Immunogenicity of a DNA-based Vaccine (COVIGEN) in Healthy Volunteers
Acronym: COVALIA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Bionet Co., Ltd (Industry); Technovalia (Industry); Telethon Kids Institute (Other); Institute for Clinical Pathology and Medical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: COV101
Record Dates: First submitted 2021-01-28; First posted 2021-02-08 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: SARS-CoV2 COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Non-blind staff preparing and administering vaccine or placebo do not participate in any other aspects of the study. Remaining trial staff and participant are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part A: Arm1 (COVIGEN (C19) 0.8 mg ID or Placebo ID) (Experimental): Participants will be randomized to receive either COVIGEN C19 (0.8 mg) given by ID (n=40) or saline placebo (n=10), administered in a two dose regimen, 28 days apart.
  Interventions: Biological: COVIGEN C19 0.8 mg ID or Placebo ID
- Part A: Arm2 (COVIGEN (C19) 2.0 mg IM or Placebo IM) (Experimental): Participants will be randomized to receive either COVIGEN C19 (2 mg) given by IM (n=40) or saline placebo (n=10), administered in a two dose regimen, 28 days apart.
  Interventions: Biological: COVIGEN C19 2.0 mg IM or Placebo IM
- Part A; Arm 3 (COVIGEN (C19) 4.0 mg IM or Placebo IM) (Experimental): Participants will be randomized to receive either COVIGEN C19 (4 mg) given by IM (n=40) or saline placebo (n=10), administered in a two dose regimen, 28 days apart
  Interventions: Biological: COVIGEN C19 4.0 mg IM or Placebo IM
- Part B: Arm 1 (COVIGEN (C20) 1.0 mg ID) in BNT162b2 primed participants (Experimental): Participants in Part B who have received a 2 dose primary course of Pfizer BNT162b2 vaccine will receive COVIGEN C20 (1mg) vaccine given by ID (n=25)
  Interventions: Biological: COVIGEN C20 1.0mg vaccine ID
- Part B: Arm 2 (COVIGEN (C20) 1.0 mg ID) in ChAdOx1-S primed participants (Experimental): Participants in Part B who have received a 2 dose primary course of Astra Zeneca ChAdOx1-S vaccine will receive COVIGEN C20 (1mg) vaccine given by ID (n=25)
  Interventions: Biological: COVIGEN C20 1.0mg vaccine ID

INTERVENTIONS:
Biological: COVIGEN C19 0.8 mg ID or Placebo ID — 2 doses of COVIGEN C19 0.8 mg ID or Placebo ID will be given at Day 1 and Day 29.
  Arms: Part A: Arm1 (COVIGEN (C19) 0.8 mg ID or Placebo ID)
Biological: COVIGEN C19 2.0 mg IM or Placebo IM — 2 doses of COVIGEN C19 2.0 mg IM or Placebo IM will be given at Day 1 and Day 29.
  Arms: Part A: Arm2 (COVIGEN (C19) 2.0 mg IM or Placebo IM)
Biological: COVIGEN C19 4.0 mg IM or Placebo IM — 2 doses of COVIGEN C19 4.0 mg IM or Placebo IM will be given at Day 1 and Day 29.
  Arms: Part A; Arm 3 (COVIGEN (C19) 4.0 mg IM or Placebo IM)
Biological: COVIGEN C20 1.0mg vaccine ID — COVIGEN C20 1.0mg ID vaccine will be given at Day 1
  Arms: Part B: Arm 1 (COVIGEN (C20) 1.0 mg ID) in BNT162b2 primed participants; Part B: Arm 2 (COVIGEN (C20) 1.0 mg ID) in ChAdOx1-S primed participants

SUMMARY:
In this trial, we are evaluating the safety and tolerability of a new investigational DNA vaccine to protect against SARS CoV-2 virus, called COVIGEN, that is developed by a company called BioNet-Asia.

A device will be used to inject the vaccine that does not require the use of a needle (needle-free injection made by a company called Pharmajet). For delivery into the skin (intradermally) a device called "Tropis" will be used, and for delivery into the muscle (intramuscularly) a device called "Stratis" will be used.

This is a 2 part study

In Part A vaccine naive participants will be given 2 vaccinations, either two active vaccines or two placebo vaccines on Day 1 and Day 29. COVIGEN C19 vaccine will be used in Part A

In Part B participants who have previously received a 2-dose primary COVID vaccine schedule will be given a booster dose of active vaccine. COVIGEN C20 vaccine will be used in Part B.

Participants in part A and B will be followed up using a combination of on-site and telephone visits for assessment of safety and immunogenicity for 12 months from 1st vaccination.

DETAILED DESCRIPTION:
Part A Vaccine Naïve participants: The study comprises three dose groups (0.8 mg COVIGEN, administered ID, 2 mg COVIGEN, administered IM and 4 mg COVIGEN, administered IM) with 50 participants in each group. Each group of 50 participants comprises two sub-groups: 25 young adults and 25 older adults. Within each group and within each sub-group, participants will be randomised 4:1 to receive COVIGEN or placebo in a double-blind fashion.

Participants will receive 2 study vaccinations, 28 days apart (Day 1 and Day 29). Each dose will be divided into 2 injections, with each injection being administered using a needle free injection system into the upper arm (left and right) at each visit.

The study will utilise a sequential dose-escalating design with a 48-hour observation period required for sentinel participants prior to the decision to dose escalate. Enrolment of the remainder of each age cohort will commence at least 48 hours after the last of the sentinel participants has received a vaccine. A Safety Review Committee (SRC) will supervise enrolment and monitoring of participant safety throughout the trial

Part B: Vaccine booster participants: The study comprises a single dose group (1.0mg COVIGEN, administered ID) to 50 participants in total, comprising 25 participants who have received a primary course of 2 doses of Pfizer BioNTech vaccine and 25 participants who have received a primary course of 2 doses of Astra Zeneca vaccine.

The dose will be divided into 2 injections, with each injection being administered using a needle free injection system into the upper arm (left and right) at each visit.

Participants will be followed up using a combination of on-site and telephone visits for assessment of safety and immunogenicity for 12 months from 1st vaccination.

ELIGIBILITY:
INCLUSION CRITERIA

Potential participants must fulfil all of the following inclusion criteria to be eligible to participate in the study:

1. Willing and capable of providing written informed consent prior to the performance of any study-specific procedure.
2. Male or female, ≥18.0 to ≤75. years of age, at the time of consent.
3. The participant must be in good health, as established by pertinent medical history, physical examination and vital signs assessments performed at Screening.
4. Body mass index (BMI) of 18 to 40 kg/m2, inclusive, at Screening.
5. Women of childbearing potential must have a negative urine pregnancy test at Screening and pre-dose on Day 1, and must agree to remain sexually abstinent, use medically effective contraception (see Section 4.3.10), or have a partner who is sterile or same-sex, from Screening until at least 90 days after the 2nd vaccination (Part A) or the Booster (Part B).

   a. Females with natural amenorrhea for <2 years (without an alternative medical cause) and who are not surgically sterile, i.e. tubal ligation, bilateral oophorectomy, or complete hysterectomy will only be considered not to be of childbearing potential if they have a documented follicle-stimulating hormone (FSH) value in the postmenopausal range.
6. Sexually active male participants who are considered sexually fertile must agree to use either a barrier method of contraception from the time of 1st vaccination until at least 90 days after the 2nd vaccination (Part A) or the Booster (Part B), or have a same sex partner, or have a partner who is permanently sterile or unable to become pregnant;
7. Both male and female participants must agree to refrain from sperm and egg donation from the day of the 1st vaccination until at least 90 days after the 2nd vaccination (Part A) or the Booster (Part B)..
8. Clinical safety laboratory evaluations at Screening must be toxicity Grade 0 or 1, or deemed not clinically significant by the Investigator.
9. The participant must agree to refrain from donating blood or plasma during the study for non-study purposes.
10. The participant must agree to have study samples retained for secondary research including exploratory analyses.
11. The participant must be able to attend all scheduled visits and to understand and comply with planned study procedures, in the Investigator's judgement.
12. Part B only: The participant must have completed a primary course (2 doses) of either Comirnaty (Pfizer BioNTech) or Astra Zeneca vaccine and ≥3 months (≥90 days) has elapsed since receipt of dose 2 in the primary course.

EXCLUSION CRITERIA

If any of the following exclusion criteria apply, the potential participant will not be permitted to participate in the study:

1. Female participant who is breastfeeding or intends to become pregnant from Screening until at least 90 days after the 2nd vaccination (Part A) or at least 90 days after booster vaccination (Part B).
2. History of any major (per Investigator's discretion) cardiovascular, renal, neurological, metabolic, gastrointestinal, hepato-biliary, uncontrolled hypertension and diabetes, clinically significant chronic pulmonary disease, asthma (with the exception of history of resolved childhood asthma), immunological and autoimmune diseases or any condition which, in the opinion of the Investigator, might interfere with the evaluation of the study objectives.
3. Chronic use (more than 14 continuous days) of systemic corticosteroids within 30 days prior to Screening. Intra-articular, intra-bursal, or topical (skin or eyes) corticosteroids are permitted.
4. History of any haematological malignancy or active neoplastic disease (excluding non-melanoma skin cancer that was successfully treated). Active is defined as having received treatment within the past 5 years.
5. History of demyelinating disease or Guillain Barre syndrome.
6. Eczema or other significant skin lesion, infection or tattoo at the site of vaccination (left or right upper arm).
7. History of blood dyscrasia or significant disorder of coagulation that, in the opinion of the Investigator, contraindicates IM injection (Part A only).
8. History of known or suspected hypersensitivity or any severe allergic reaction including anaphylaxis, generalised urticaria, angioedema, and other significant reaction to Kanamycin or any vaccine component,.
9. Presence of active viral or bacterial infection, with or without fever (oral temperature ≥37.8 °C) at Screening or within 72 hours prior to each vaccination, if determined by the Investigator to be of clinical significance (enrolment [provided Screening period does not exceed 30 days] or dosing may be delayed for full recovery if acceptable to the Investigator).
10. Positive serological test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody or HIV (Type 1 or 2) antibody at Screening.
11. Known current or previous laboratory confirmed SARS-CoV-2 infection/COVID 19, or positive for SARS-CoV-2 infection, either by SARS CoV 2-specific IgG antibody (Part A only) or RT-PCR, at Screening.
12. Suspected SARS-CoV-2 infection/COVID-19, including individuals who are required to self-isolate.
13. Individuals currently working in occupations with high risk of exposure to SARS CoV-2, e.g. healthcare workers in direct care of COVID-19 patients, emergency responders or front-line workers.
14. Receipt of any other SARS-CoV-2 or other experimental coronavirus vaccine at any time prior to the study or planned receipt of any other SARS-CoV-2 or other experimental vaccine within 57 days of receipt of the 1st study vaccination (Part A only).
15. Receipt of any other experimental coronavirus vaccine at any time prior to the study or planned receipt of any other SARS-CoV-2 or other experimental vaccine within 29 days of receipt of the booster vaccination (Part B only).
16. Participating in any other clinical study and have received any other investigational product (i.e. study vaccine, drug, biologic or device) within 30 days or 5 half-lives (whichever is longer) prior to Screening, or are taking part in a non medication study which, in the opinion of the Investigator, would interfere with the interpretation of the assessments in this study.
17. Received or plans to receive a live-attenuated vaccine within 4 weeks before or after each study vaccination.
18. Received or plans to receive an inactivated vaccine within 2 weeks before or after each study vaccination (including influenza vaccines).
19. Received immunoglobulins and/or any blood or blood products within 3 months before the 1st vaccination (Part A) or before the booster vaccination (Part B) or plans to receive any blood or blood products at any time during the study.
20. Has a history of alcohol abuse, or other drug abuse assessed as a dependency problem by the Investigator within 6 months before the 1st vaccination (Part A) or before the booster vaccination (Part B).
21. Has any psychiatric or cognitive disease that, in the opinion of the Investigator, may interfere with the participant's ability to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Frequency of solicited local reactogenicity AEs | Through 7 days after each vaccination (Day 1, 29 for Part A and Day 1 for Part B)
  Percentage of participants with any local reaction (pain, swelling/induration, erythema/redness) for 7 days following each vaccination
Frequency of solicited systemic reactogenicity AEs | Through 7 days after each vaccination (Day 1, 29 for Part A and Day 1 for Part B)
  Percentage of participants with any systemic reaction (fever, fatigue, chills, myalgia, arthralgia, headache, nausea/vomiting and diarrhea) for 7 days following each vaccination
Frequency of any unsolicited AEs | Day 1 to Day 57 after the 1st vaccination (Part A) or from Day 1 to Day 29 after booster vaccination (Part B).
  Percentage of participants with unsolicited AEs up to Day 57
Frequency of any serious adverse events (SAEs) | Day 1 to 12 months after 1st vaccination
  Percentage of participants with SAEs from Day 1 to 12 months after 1st vaccination
Frequency of any medically attended adverse events (MAAES) | From Day 1 to 12 months after the 1st vaccination
  Measured by MedDRA classification, severity score and relatedness.
Change in safety laboratory values from baseline | From Day1 to Day 36 in Part A and from Day 1 to Day 8 in Part B
  Number of participants with abnormal laboratory values (haematology, chemistry and urinalysis) by FDA toxicity scoring.

SECONDARY OUTCOMES:
GMTs for serum neutralizing antibody response | At day1, day 29 and day 57 (Part A) and Day 1, Day 8, Day 29 (Part B only);
  Level of neutralizing antibodies as measured by SARS-CoV-2 Neutralization assay
GMFR from baseline for serum neutralizing antibody response | At day 57 (Part A) or day 29 (Part B)
  Measured by SARS-CoV-2 Neutralization assay
Seroconversion rate for serum neutralizing antibody response | At day 57 compare to baseline for Part A and at day 29 compare to baseline for Part B
  Defined as proportion of participants with a with a ≥4-fold rise
GMTs for serum S1- and RBD-specific IgG antibody responses | At day 1, day 29 and day 57 (Part A) and at Day 1, Day 8, Day 29; (Part B only)
  SARS-CoV-2 anti-S1 and anti-RBD IgG antibody ELISAs
GMFR from baseline for serum S1- and RBD-specific IgG antibody responses | At day 57 (Part A) and at day 29 (Part B)
  As measured by ELISA
Seroconversion rate serum S1- and RBD-specific IgG antibody responses | At day 57 compare to baseline for Part A and at day 29 compare to baseline for Part B
  Defined as the proportion of participants with a ≥ 4-fold rise
Geometric means of T-cells (spot-forming cells) producing IFNγ, IL-2, or both for S protein specific IFN-γ and IL-2 T-cell responses | At day 1, day 29, and day 57 (Part A) or at Day 1, Day 8, and Day 29 (Part B only)
  SARS-CoV-2 Spike Protein dual IFN-γ and IL-2 T-cell ELISpot (FluoroSpot)
Fold rise of T-cells (spot-forming cells) producing IFNγ, IL-2, or both for S protein specific IFN-γ and IL-2 T-cell responses | At day 57 compared to baseline for Part A and at day 29 compare to baseline for Part B
  SARS-CoV-2 Spike Protein dual IFN-γ and IL-2 T-cell ELISpot (FluoroSpot)
Proportion of participants with significant T-cell responses for S protein specific IFN-γ and IL-2 T-cell responses | At day 57 for Part A and at day 29 for Part B
  IL-2 T-cell ELISpot (FluoroSpot)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas WOOD, MB BS FRACP PhD., Principal Investigator — University of Sydney
Locations (3):
- Australia (3):
  - Scientia Clinical Research, Randwick, New South Wales
  - Vaccinology and Immunology Research Trials Unit, Women's and Children's Hospital, Adelaide, South Australia
  - Wesfarmers Centre of Vaccines and Infectious Diseases Telethon Kids Institute, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Undecided